CLINICAL TRIAL: NCT01946529
Title: Therapeutic Trial for Patients With Ewing Sarcoma Family of Tumor and Desmoplastic Small Round Cell Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Tennessee (Other); University of Florida (Other); Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESFT13; NCI-2013-01657 (Registry Identifier: NCi Clinical Trial Registration Program)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2016-10-19 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Desmoplastic Small Round Cell Tumor; Ewing Sarcoma of Bone or Soft Tissue; Localized Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Vincristine; Doxorubicin; Cyclophosphamide; Ifosfamide; Etoposide; Temozolomide; temsirolimus; Bevacizumab; Sorafenib; Surgical Procedures, Operative; Radiation; Proton Therapy; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Standard Risk) (Active Comparator): Participants will receive vincristine, doxorubicin, cyclophosphamide, ifosfamide and etoposide. Doxorubicin will be omitted following a total cumulative dose of 375 mg/m^2. Depending on the size and location of the participant's tumor, they will have surgery alone, radiation alone, or surgery followed by radiation. Local control measures (surgery and/or radiation therapy) will be instituted after 6 courses of chemotherapy. Total duration of treatment is approximately 29 weeks.
  Interventions: Drug: vincristine; Drug: doxorubicin; Drug: cyclophosphamide; Drug: ifosfamide; Drug: etoposide; Procedure: surgery; Radiation: radiation
- Group B (High Risk) (Active Comparator): Participants will receive vincristine, doxorubicin, cyclophosphamide, ifosfamide, etoposide, irinotecan, temozolomide, temsirolimus, bevacizumab, and sorafenib. Depending on the size and location of the participant's tumor, they will have surgery alone, radiation alone or surgery followed by radiation.
  Interventions: Drug: doxorubicin; Drug: cyclophosphamide; Drug: ifosfamide; Drug: etoposide; Drug: temozolomide; Drug: temsirolimus; Drug: bevacizumab; Drug: sorafenib; Procedure: surgery; Radiation: radiation

INTERVENTIONS:
Drug: vincristine — Dosage and route of administration: Infants < 12 months of age: 0.05 mg/kg IV day 1; participants ≥ 12 months of age: 1.5 mg/m^2 IV day 1 (max. dose 2 mg).
  Other Names: Oncovin(R)
  Arms: Group A (Standard Risk)
Drug: doxorubicin — Dosage and route of administration: Infants < 1 year 2.5 mg/kg continuous infusion (CI) over 48 hours, days 1-2; participants > 1 year of age 75 mg/m^2 CI over 48 hours, days 1-2.
  Other Names: Adriamycin(R)
Drug: cyclophosphamide — Dosage and route of administration: The dose and route are different in neo-adjuvant/adjuvant chemotherapy and maintenance therapy. Please see the Detailed Description for further information.
  Other Names: Cytoxan(R)
Drug: ifosfamide — Dosage and route of administration: Infants < 1 year of age 60 mg/kg/day IV over 60 minutes days 1-5; participants > 12 months of age 1800 mg/m^2 IV over 60 minutes x 5 days, days 1-5.
  Other Names: Ifex(R)
Drug: etoposide — Dosage and route of administration: Infants < 1 year of age 3.3 mg/kg/day IV over 60 minutes days 1-5; children > 1 year 100 mg/m^2 daily IV over 60 minutes days 1-5.
  Other Names: VP-16; Vepesid(R)
Drug: temozolomide — Dosage and route of administration: Temozolomide 100 mg/m^2 PO once daily, days 1-5.
  Other Names: Temodar(R)
  Arms: Group B (High Risk)
Drug: temsirolimus — Dosage and route of administration: Temsirolimus 35 mg/m^2 IV once day 1 and day 8.
  Other Names: CCI-779; Torisel^TM
  Arms: Group B (High Risk)
Drug: bevacizumab — Dosage and route of administration: Bevacizumab 15 mg/kg IV on day 1 every 3 weeks.
  Other Names: rhumab VEGF; Avastin(R)
  Arms: Group B (High Risk)
Drug: sorafenib — Dosage and route of administration: 90 mg/m^2/dose PO BID
  Other Names: BAY-43-9006; Nexavar(R)
  Arms: Group B (High Risk)
Procedure: surgery — If participant meets the criteria, they will have surgical resection of their tumor.
  Other Names: therapeutic conventional surgery
Radiation: radiation — If the participant meets the criteria, participants will receive radiation therapy. Chemotherapy will continue during radiation.
  Other Names: proton beam radiation therapy; external beam radiation therapy; brachytherapy

SUMMARY:
This protocol will study treatment for Ewing sarcoma family of tumors (ESFT) and desmoplastic small round cell tumor (DSRCT). Participants with ESFT will be divided into two treatment groups, A or B, based on tumor characteristics.

Group A (standard risk) participants have tumor that is not in the pelvis, has not spread to other parts of the body, and are less than 14 years of age. Because previous clinical trials have shown that standard treatment is very effective for children whose tumors have these characteristics, these participants will receive standard treatment.

Group B (high risk) participants are 14 years of age or older or have tumor in the pelvis, or the tumor has spread to other parts of the body. Participants with DSRCT in the abdomen and/or pelvis or with tumor that cannot be removed by surgery alone or has spread to other parts of the body will be included in Group B. Participants in this group are considered high risk because there is a greater chance of tumor recurring following standard treatments currently in use.

All participants will be followed and evaluated for 10 years following completion of therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

* To estimate the response rate to two initial courses of temsirolimus, temozolomide and irinotecan in previously untreated patients with high-risk Ewing sarcoma family of tumors (ESFT).

SECONDARY OBJECTIVES:

* To estimate the overall survival and progression-free survival in participants with ESFT treated with these approaches.
* To estimate the time to progression in participants with ESFT treated in Group B (high risk).
* To estimate the cumulative incidence of local failure following local control paradigm in this trial.

Group A:

Participants will receive interval compressed (every 2 weeks) alternating courses of chemotherapy with vincristine, doxorubicin, and cyclophosphamide (VDC) and with ifosfamide and etoposide (IE). Doxorubicin will be omitted following a total cumulative dose of 375 mg/m^2. Local control measures (surgery and/or radiation therapy) will be instituted after 6 courses of chemotherapy. Total duration of treatment is approximately 29 weeks.

Group B:

Participants eligible for the window therapy will receive two courses (21 days duration each) of mTOR inhibitor, temsirolimus, in combination with temozolomide and irinotecan. Irinotecan (20 mg/m^2) will be administered IV on a protracted schedule of daily for 5 days, 2 days off, repeated daily x 5 [(qdx5)x2], temozolomide (100 mg/m^2) PO daily x 5 days and temsirolimus 35 mg/m^2 IV weekly on day 1 and 8. Following window treatment (weeks 1 - 6), participants will proceed to induction chemotherapy (weeks 7 - 33) consisting of interval compressed (every 2 weeks) alternating courses of chemotherapy with vincristine, doxorubicin, and cyclophosphamide (VDC) with ifosfamide and etoposide (IE). Doxorubicin will be omitted following a total cumulative dose of 375 mg/m^2. Local control measures (surgery and/or radiation therapy) will be instituted after 6 courses of induction chemotherapy (week 19). Participants whose tumors respond to window therapy will receive temsirolimus, temozolomide and irinotecan at weeks 29 and 31 in place of ifosfamide and etoposide. Following induction therapy, participants will receive six 21-day courses of maintenance therapy consisting of bevacizumab IV on day 1 and daily oral sorafenib and low-dose cyclophosphamide day 1 through day 21.

ELIGIBILITY:
Inclusion Criteria:

* Group A participants must be <14 years of age at time of diagnosis of histologically proven non-pelvic localized Ewing sarcoma family of tumor (ESFT) involving the bone or soft tissue.
* Group B participants must have newly diagnosed of histologically proven ESFT involving the bone or soft tissue and at least one of the following: metastatic disease (must be biopsy proven), or pelvic primary, or ≥14 years of age at the time of diagnosis.
* OR Group B participants must be newly diagnosed with intra-abdominal, unresectable or metastatic desmoplastic small round cell tumor. Metastatic site must be biopsy proven.
* Age must be ≤25 years.
* Adequate bone marrow function defined as a peripheral absolute neutrophil count (ANC) ≥750/m^3 and platelet count ≥75,000/m^3 (no transfusion within 7 days of study enrollment). Patients with Ewing sarcoma metastatic to the bone marrow are not required to meet bone marrow criteria for study eligibility and are not evaluable for hematologic toxicity.
* Must have adequate renal function based on age.
* Must not have had prior chemotherapy or radiation therapy. Emergent radiotherapy to preserve vital organ function is permitted. Participants who receive emergent radiation will not be eligible for window therapy.
* Must have adequate hepatic function defined as total bilirubin ≤3.0 mg/dL.
* Must have adequate cardiac function defined as shortening fraction ≥28%.
* Females of childbearing potential and males able to father a child must be willing to practice acceptable methods of birth control to prevent pregnancy.
* Additional criteria for Group B participants who will receive upfront window therapy (does not apply to participants who opt out of window therapy):

  * Cytochrome P450 CYP3A4 active agents: Must not be taking any of the following potent CYP3A4 inducers or inhibitors within 1 week prior to study entry: azole antifungals (such as fluconazole, voriconazole, itraconazole, ketoconazole), rifampin, phenytoin, phenobarbitol, carbamazepine, grapefruit juice and St. John's wort.
  * Must have measurable disease.
  * Must not have received emergent radiation therapy.
  * Serum triglyceride level ≤ 300 mg/dL and serum cholesterol ≤ 300 mg/dL.
  * Random or fasting glucose within the upper limits of normal for age. If random glucose is elevated, fasting glucose must be within normal range.
  * SGOT (AST) and SGPT (ALT) ≤3.0 x upper limit of normal for age.

Exclusion Criteria:

* Participant is pregnant or breastfeeding.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Participant has a prior history of malignancy, with the exception of non-melanoma skin cancer. Participants with history of skin cancer must have 5 years elapse since that diagnosis, be in remission, and must not have received chemotherapy, immunotherapy, or radiation therapy.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12-27 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sara M. Federico, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at St. Jude Children's Research Hospital between December 2013 and June 2015.
Groups:
- Group B (High Risk) - ESFT: Group B participants with a diagnosis of Ewing Sarcoma Family of Tumor (ESFT).
- Group B (High Risk) - DSRCT: Group B participants with a diagnosis of Desmoplastic Small Round Cell Tumor (DSRCT).
Period: End of Window Therapy (2 Courses)
Arm/Group | Group A (Standard Risk) | Group B (High Risk) - ESFT | Group B (High Risk) - DSRCT
Started | 1 | 17 | 6
Completed | 1 | 16 | 6
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Completion of All Therapy
Arm/Group | Group A (Standard Risk) | Group B (High Risk) - ESFT | Group B (High Risk) - DSRCT
Started | 1 | 16 | 6
Completed | 0 | 0 | 0
Not Completed | 1 | 16 | 6
Not completed — Some pts. still receiving study therapy | 1 | 16 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Standard Risk) | Group B (High Risk) - ESFT | Group B (High Risk) - DSRCT | Total
Number analyzed (Participants) | 1 | 16 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (0) | 13.0 (5.7) | 14.7 (4.1) | 13.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 9 | 1 | 10
  Male | 1 | 7 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 1 | 14 | 3 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Primary disease site [Number; unit: participants]
  Pelvis | 0 | 6 | 5 | 11
  Other | 1 | 10 | 1 | 12
Disease stage [Number; unit: participants]
  Metastases | 0 | 11 | 5 | 16
  Local | 1 | 5 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Response to Window Therapy (2 Courses) for Group B (High-risk) - ESFT Participants
Description: Response rate will be defined as the proportion of patients who achieved complete response or partial response (CR+PR) using the World Health Organization (WHO) criteria evaluated after two initial courses of temsirolimus, temozolomide and irinotecan in previously untreated patients with high risk Ewing Sarcoma Family of Tumor (ESFT). Participants who are treated in Group B with Desmoplastic Small Round Cell Tumor (DSRCT) or those who do not receive window therapy will not be included in this analysis.
Time Frame: at 6 weeks after start of therapy (after 2 initial courses)
Population: Of the 17 Group B participants with high-risk ESFT, 12 received window therapy and are considered evaluable for this outcome.
Measure: Number; unit: participants
Groups:
- Group B (High Risk) - ESFT: Participants received vincristine, doxorubicin, cyclophosphamide, ifosfamide, and etoposide. Patients with measurable disease were eligible to receive irinotecan, temozolomide, and temsirolimus. Additionally, all patients were eligible to receive a maintenance therapy at the end of treatment including bevacizumab and sorafenib. Depending on the size and location of the participant's tumor, they had surgery alone, radiation alone, or surgery followed by radiation.
Arm/Group | Group B (High Risk) - ESFT
Number analyzed (Participants) | 12
participants
  Partial Response (PR) | 3
  Stable disease (no response) (NR) | 8
  Progressive Disease (PD) | 1

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time interval from the date on study to the date of death or the date of last follow-up. OS will be estimated using the method of Kaplan-Meier for group A and B participants, respectively.
Time Frame: Maximum of 11 years after the start of therapy
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time interval from the date on study to the date of disease progression or death or the date if last follow-up. PFS will be estimated using the method of Kaplan-Meier for group A and B participants, respectively.
Time Frame: Maximum of 11 years after the start of therapy
Reporting Status: Not Posted

4. Secondary Outcome: Time to Progression
Description: Median time to progression of group B patients will be estimated from the Kaplan-Meier curve.
Time Frame: Maximum of 11 years after the start of therapy
Reporting Status: Not Posted

5. Secondary Outcome: Local Failure Rate
Description: Loco-regional failure is defined as the time interval from date of start of local therapy to date of loco-regional failure. Distant failure or death prior to loco-regional failure will be considered competing events in the analyses. The cumulative incidence of loco-regional failure will be estimated using methods described in Kalbfleisch and Prentice.
Time Frame: Maximum of 11 years after the start of therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the on-study date through 05/03/2016.
Groups:
- Group B (High Risk) - Total: All Group B High Risk participants with ESFT or DSRCT.
  Participants received vincristine, doxorubicin, cyclophosphamide, ifosfamide, and etoposide. Patients with measurable disease were eligible to receive irinotecan, temozolomide, and temsirolimus. Additionally, all patients were eligible to receive a maintenance therapy at the end of treatment including bevacizumab and sorafenib. Depending on the size and location of the participant's tumor, they had surgery alone, radiation alone, or surgery followed by radiation.
Arm/Group | Group A (Standard Risk) | Group B (High Risk) - ESFT | Group B (High Risk) - DSRCT | Group B (High Risk) - Total
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/16 | 0/6 | 1/22
Other Adverse Events (participants affected / at risk) | 1/1 | 16/16 | 6/6 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Standard Risk) (N=1) | Group B (High Risk) - ESFT (N=16) | Group B (High Risk) - DSRCT (N=6) | Group B (High Risk) - Total (N=22)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Standard Risk) (N=1) | Group B (High Risk) - ESFT (N=16) | Group B (High Risk) - DSRCT (N=6) | Group B (High Risk) - Total (N=22)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 15 (66) | 6 (21) | 21 (87)
Lymphocyte count decreased (Investigations) | 1 (7) | 15 (215) | 6 (48) | 21 (263)
Neutrophil count decreased (Investigations) | 1 (6) | 15 (133) | 6 (36) | 21 (169)
White blood cell decreased (Investigations) | 1 (4) | 15 (150) | 6 (36) | 21 (186)
Hypertension (Vascular disorders) | 1 (6) | 11 (60) | 5 (22) | 16 (82)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 9 (22) | 3 (4) | 12 (26)
Anemia (Blood and lymphatic system disorders) | 1 (3) | 16 (96) | 6 (34) | 22 (130)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 15 (130) | 6 (32) | 21 (162)
Weight loss (Investigations) | 0 (0) | 13 (33) | 5 (12) | 18 (45)
Vomiting (Gastrointestinal disorders) | 0 (0) | 12 (51) | 5 (19) | 17 (70)
Platelet count decreased (Investigations) | 0 (0) | 12 (41) | 5 (7) | 17 (48)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 11 (31) | 4 (10) | 15 (41)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 11 (33) | 4 (6) | 15 (39)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 10 (19) | 4 (10) | 14 (29)
Nausea (Gastrointestinal disorders) | 0 (0) | 10 (35) | 4 (7) | 14 (42)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (32) | 2 (3) | 14 (35)
Proteinuria (Renal and urinary disorders) | 0 (0) | 9 (23) | 4 (8) | 13 (31)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 10 (15) | 2 (2) | 12 (17)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 10 (19) | 2 (4) | 12 (23)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 9 (24) | 3 (13) | 12 (37)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 9 (38) | 2 (2) | 11 (40)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 8 (10) | 2 (4) | 10 (14)
Fatigue (General disorders) | 0 (0) | 7 (7) | 3 (4) | 10 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 8 (30) | 2 (5) | 10 (35)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 7 (27) | 2 (4) | 9 (31)
Fever (General disorders) | 0 (0) | 7 (12) | 1 (3) | 8 (15)
Allergic reaction (Immune system disorders) | 0 (0) | 6 (6) | 2 (3) | 8 (9)
Constipation (Gastrointestinal disorders) | 0 (0) | 7 (8) | 0 (0) | 7 (8)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (13) | 2 (3) | 7 (16)
Colitis (Gastrointestinal disorders) | 0 (0) | 5 (6) | 1 (1) | 6 (7)
Mucosa infection (Infections and infestations) | 0 (0) | 5 (6) | 1 (1) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (8) | 2 (3) | 6 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 5 (40) | 1 (5) | 6 (45)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 1 (1) | 6 (7)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (2) | 5 (6)
Hematuria (Renal and urinary disorders) | 0 (0) | 4 (7) | 1 (1) | 5 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (1) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 4 (8) | 0 (0) | 4 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (7) | 1 (1) | 4 (8)
Malaise (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 3 (5) | 0 (0) | 3 (5)
Lung infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
GGT increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Esophageal infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Cardiac troponin T increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (4)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 1 (1) | 2 (4)

LIMITATIONS AND CAVEATS:
Interim analysis to evaluate efficacy of the therapy determined that the window therapy did not meet the anticipated response, and trial accrual was stopped. Some patients continue on therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes